CLINICAL TRIAL: NCT06978673
Title: Comparison of Neurolytic Block Techniques for the Treatment of Abdominal Visceral Pain and Their Influence On The Quality of Life of Patients With Cancer
Brief Title: Neurolytic Block Techniques In Abdominal Visceral Cancer Pain
Acronym: CONCERN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, amsousa, Coordinator of the Pain Group at the Instituto do Cancer do Estado de São Paulo., Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NP 076-210
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cancer, Malignant Tumors; Abdominal Cancer; Cancer Pain; Visceral Pain; Cancer-related Pain; Pain Management; Celiac Ganglia; Sympathetic Ganglia
Keywords: cancer pain; visceral pain; abdominal cancer; cancer; abdominal pain; cancer-related pain; pain management; neurolytic block; splanchnic nerve block; celiac plexus block; sympathetic neurolysis
MeSH Terms: conditions — Neoplasms; Cancer Pain; Visceral Pain; Agnosia; Abdominal Pain | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CELIAC PLEXUS NEUROLYSIS (Active Comparator): The patient, under sedation and breathing spontaneously with oxygen support, will be placed in the horizontal prone position. Fluoroscopy will be used to locate the first lumbar vertebra, which will serve as a reference for the puncture site. Two 22G × 15 cm needles will be introduced bilaterally, up to 6 cm from the midline at the level of L1, and directed superiorly toward the transverse process of L1 under coaxial vision. Once they reach the vertebral body bilaterally, the needles will be positioned anterior to the vertebral body of L1, in the retroperitoneal region. The needle stylet will be removed, and the absence of blood, cerebrospinal fluid, or urine returning through the needle will be verified. If none of these signs are present, 2 ml of non-ionic contrast will be administered through the needle to confirm proper positioning in the retroperitoneum. After confirmation, 5 ml of absolute alcohol will be injected bilaterally.
  Interventions: Procedure: Celiac Plexus Neurolysis - 5 ml of absolute alcohol (100%)
- SPLANCHNIC NERVE NEUROLYSIS (Experimental): The patient, under spontaneous breathing with oxygen support, will be placed in the horizontal prone position and supported by cushions placed under the iliac crests and chest. With a mark maintained over T11, the fluoroscopy machine will be positioned obliquely (approximately 45º), and the movement of the diaphragm-as well as its relationship with the vertebral body-will be observed during inspiration and expiration. The entry point will be at the junction of the rib and the vertebral body. The needle will be introduced using coaxial visualization to reach the lateral aspect of the vertebral body, near the costovertebral angle. With the fluoroscopy in profile, the needle will be advanced to the anterior third of the vertebral body, and any return of blood or cerebrospinal fluid will be checked. Non-ionic contrast will then be injected to confirm the needle position in both anteroposterior and lateral views. Finally, 5 ml of absolute alcohol will be injected through each needle.
  Interventions: Procedure: Splanchnic nerve neurolysis - 5 ml of absolute alcohol (100%)

INTERVENTIONS:
Procedure: Splanchnic nerve neurolysis - 5 ml of absolute alcohol (100%) — Splanchnic neurolysis will be performed with 5 ml of absolute alcohol on each side at the level of the eleventh thoracic vertebra.
  Other Names: SPLANCHNIC NERVE BLOCK; SPLANCHNIC NERVE BLOCKADE; SPLANCHNIC BLOCK
  Arms: SPLANCHNIC NERVE NEUROLYSIS
Procedure: Celiac Plexus Neurolysis - 5 ml of absolute alcohol (100%) — Celiac plexus neurolysis will be performed with 5 ml of absolute alcohol on each side at the level of the first lumbar vertebra.
  Other Names: Celiac plexus block
  Arms: CELIAC PLEXUS NEUROLYSIS

SUMMARY:
The neurolytic blocks of sympathetic chains are commonly used for the treatment of cancer-related pain. This study aims to compare celiac plexus neurolysis and splanchnic nerve neurolysis for the treatment of abdominal visceral pain and its influence on the quality of life of patients with cancer.

DETAILED DESCRIPTION:
Double-blind randomized clinical trial.

The objective of the study is to compare the analgesic efficacy of splanchnic nerve neurolysis with alcohol to celiac plexus block with alcohol, with pain relief as the primary outcome. It also aims to quantify the adverse effects of the techniques as secondary outcomes. The sample size calculation will be based on comparing the mean pain scores on the Numerical Rating Scale of patients in the Control Group and the Intervention Group, evaluated after completing the second month of treatment. A two-tailed t-test will be sufficient and will require an adequate sample size. Therefore, for the chosen sample design with a significance level of α=5%, a power of 1-β=80%, assuming M1=5.0 and M2=3.5 and a standard deviation of 2.0, the sample size required is n=58. the sample size required is n=58. Considering a 10% dropout rate, the final sample size will be increased to 64 participants. Convenience sampling (a non-probabilistic sampling method) will be used. Participants will be randomly allocated to the groups using a list generated by a program obtained at https://www.randomizer.org. The proportion between the participants in the groups will be 1:1, with 32 patients allocated to the Intervention arm and 32 to the Control arm. The allocation of the total 64 participants will be determined by randomly assigned sequential letters (A or B) generated by the computer (website https://www.randomizer.org), randomly assigning numbers from 0 to 64 to each group: Control Group (Celiac Block) and Intervention Group (Splanchnic Nerve Block). The Control Group will receive celiac plexus neurolysis with absolute alcohol, and the Intervention Group will receive splanchnic nerve neurolysis with alcohol. The statistical analysis will be performed in program R version 3.5.1. The results obtained will be presented as mean + standard deviation for continuous data or absolute frequency for described data. For quantitative variables, the Student's t-test will be used for normally distributed data, or the Mann-Whitney test for non-normally distributed data. For qualitative variables, the chi-square test will be used or Fisher's exact test. Significant difference is defined as p < 0.05. Data will be collected and managed using REDCap data capture tools.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older Presence of localized visceral pain in the upper abdomen originating from cancer of the stomach, duodenum, distal esophagus, ascending or transverse colon, liver, biliary tract, or pancreas

Ineffectiveness of analgesic treatment with third-step opioids according to the WHO analgesic ladder, including:

Opioids (≥ 60 mg/day of morphine equivalents) Antidepressants (tricyclic or dual-action), at any dosage Gabapentinoids, at any dosage Presence of side effects from analgesics that are difficult to manage with medication

Exclusion Criteria:

Presence of ascites Presence of deep vein thrombosis Presence of hepatic failure: Child-Pugh class B or C Presence of renal failure: estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m² Use of any anticoagulant medication

Clinical coagulation disorder, defined as:

INR > 1.5 Prothrombin activity < 70% or prothrombin time > 13.5 seconds aPTT > 40 seconds Cardiovascular failure: NYHA class III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PAIN SCORE | 1st Day Post-procedure; 15th Day Post-procedure; 30th Day Post-procedure; 2nd Month Post-procedure
  Pain will be assessed using the Numerical Rating Scale (NRS), a scale from 0 to 10 where: 0 indicates no pain and 10 indicates the worst possible pain.
  Scores are typically categorized as:
  Mild pain: 0-3 Moderate pain: 4-6 Severe pain: 7-10
  Additionally, the Descriptive Verbal Scale will be used, with the following categories:
  No pain Mild pain Moderate pain Severe pain.

SECONDARY OUTCOMES:
Quality of life assessment. | 1st Day Post-procedure; 15th Day Post-procedure; 30th Day Post-procedure; 2nd Month Post-procedure
  Quality of life will be assessed using the Brief Pain Inventory - Short Form (SF-36) questionnaire, which evaluates both pain intensity and its impact on daily functioning.
  The questionnaire covers two main areas:
  Pain Severity - Patients rate their pain at its:
  Worst Least Average Current (right now) (using a 0-10 numeric scale, where 0 = no pain and 10 = pain as bad as you can imagine).
  Pain Interference - Assesses how much pain interferes with:
  General activity Mood Walking ability Normal work Relationships with others Sleep Enjoyment of life (also rated on a 0-10 scale, where 0 = does not interfere and 10 = completely interferes).
  Additionally, the questionnaire includes:
  A pain location diagram Information about current pain medications and their effectiveness Description of pain relief methods.
Adverse Events | 1st Day Post-procedure; 15th Day Post-procedure; 30th Day Post-procedure; 2nd Month Post-procedure
  Adverse events inherent to the studied procedures will be assessed and recorded. These include:
  Abdominal pain; Diarrhea; Hypotension (low blood pressure); Back pain; Nausea and vomiting; Fever; Bloating or abdominal distention; Delayed gastric emptying; Injury to surrounding structures (e.g., blood vessels or organs); Nerve damage; Impaired digestive function; Local infection at the puncture site; Loss of autonomic function; Pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Sousa, MD. PhD., Study Director — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto de Cancer Do Estado, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Koyyalagunta D, Engle MP, Yu J, Feng L, Novy DM. The Effectiveness of Alcohol Versus Phenol Based Splanchnic Nerve Neurolysis for the Treatment of Intra-Abdominal Cancer Pain. Pain Physician. 2016 May;19(4):281-92. PMID 27228515
- [Background] Ahmed A, Arora D. Fluoroscopy-guided Neurolytic Splanchnic Nerve Block for Intractable Pain from Upper Abdominal Malignancies in Patients with Distorted Celiac Axis Anatomy: An Effective Alternative to Celiac Plexus Neurolysis - A Retrospective Study. Indian J Palliat Care. 2017 Jul-Sep;23(3):274-281. doi: 10.4103/IJPC.IJPC_28_17. PMID 28827930
- [Background] Uehara Y, Matsumoto Y, Kosugi T, Sone M, Nakamura N, Mizushima A, Miyashita M, Morita T, Yamaguchi T, Satomi E. Availability of and factors related to interventional procedures for refractory pain in patients with cancer: a nationwide survey. BMC Palliat Care. 2022 Sep 26;21(1):166. doi: 10.1186/s12904-022-01056-6. PMID 36154936
- [Background] Hochberg U, Ingelmo P, Sole E, Miro J, Rivera G, Perez J. Early Interventional Treatments for Patients with Cancer Pain: A Narrative Review. J Pain Res. 2023 May 18;16:1663-1671. doi: 10.2147/JPR.S405808. eCollection 2023. PMID 37223437
- [Background] Noble M, Gress FG. Techniques and results of neurolysis for chronic pancreatitis and pancreatic cancer pain. Curr Gastroenterol Rep. 2006 Apr;8(2):99-103. doi: 10.1007/s11894-006-0004-x. PMID 16533471
- [Background] Comlek S. Pain Control with Splanchnic Neurolysis in Pancreatic Cancer Patients Unresponsive to Celiac Plexus Neurolysis. J Pain Res. 2020 Aug 12;13:2023-2031. doi: 10.2147/JPR.S266689. eCollection 2020. PMID 32848449
- [Background] Yamamuro M, Kusaka K, Kato M, Takahashi M. Celiac plexus block in cancer pain management. Tohoku J Exp Med. 2000 Sep;192(1):1-18. doi: 10.1620/tjem.192.1. PMID 11128864
- [Background] Paul A, Borkar A. Fluoroscopy-Guided Splanchnic Nerve Block for Cancer-Associated Pain. Cureus. 2022 Oct 31;14(10):e30944. doi: 10.7759/cureus.30944. eCollection 2022 Oct. PMID 36465781
- [Background] Lu F, Li X, Song L, Ye L, Wang X, Wang R. Efficacy and Safety of Celiac Plexus Neurolysis Versus Splanchnic Nerve Neurolysis in the Management of Abdominal Cancer Pain: A Meta-analysis of 359 Patients. Pain Physician. 2024 Jan;27(1):1-10. PMID 38285023